CLINICAL TRIAL: NCT06876766
Title: Effect of Pediatric Lung Ultrasound on Antibiotic Prescriptions in Hospitalized Children and Adolescents With Lower Respiratory Tract Infections.
Brief Title: Effect of Pediatric Lung Ultrasound on Antibiotic Prescriptions in Hospitalized Children and Adolescents With Lower Respiratory Tract Infections. A Randomized Controlled Trial.
Acronym: PLUS-AP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BIO-2024-0304
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Lower Resp Tract Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung Ultrasound ''LUS'' (Experimental): Participants in this group will undergo a lung ultrasound within 24 hours of enrollment. The results of this ultrasound will be used to help guide decisions about when to stop antibiotic therapy, aiming to reduce unnecessary antibiotic use.
  Interventions: Device: Lung Ultrasound
- Sham lung ultrasound ''SLUS'' (Sham Comparator): Participants in this group will receive the standard clinical care for lower respiratory tract infections, which may include diagnostic tests such as chest X-ray, with antibiotic therapy managed according to the usual clinical protocols.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Lung Ultrasound — Lung ultrasound (LUS) is a non-invasive, radiation-free imaging technique that uses sound waves to visualize the lungs. It will be used in the experimental arm to help guide decisions regarding antibiotic therapy in hospitalized children and adolescents with lower respiratory tract infections (LRTIs). The LUS will be performed within 24 hours of enrollment.
  Arms: Lung Ultrasound ''LUS''
Device: Sham — In the sham group, participants will undergo a mock or placebo version of the lung ultrasound. This involves performing the procedure in a way that mimics the real ultrasound process but does not provide any diagnostic results or influence clinical decision-making regarding antibiotic therapy.
  Arms: Sham lung ultrasound ''SLUS''

SUMMARY:
Title: Effect of Pediatric Lung Ultrasound on Antibiotic Prescriptions in Hospitalized Children and Adolescents with Lower Respiratory Tract Infections (PLUS-AP Trial)

Purpose of the Study:

This study is being done to find out if a type of imaging called lung ultrasound (LUS) can help doctors decide when to stop antibiotics in children and teens who are in the hospital with lung infections, like pneumonia. Antibiotics are often given to these patients, but sometimes they are used for longer than necessary, which can be harmful. The investigators want to see if using LUS helps doctors make decisions that reduce unnecessary antibiotic use, which can help prevent antibiotic resistance and other complications.

What is Lung Ultrasound (LUS)? Lung ultrasound is a safe, non-invasive, and painless test that uses sound waves to look at the lungs. It doesn't involve radiation like chest X-rays. It is already being used to help doctors understand lung conditions, and this study will test if it can also help in deciding when to stop antibiotics.

How the Study Works:

Participants: Children and adolescents (ages 3 months-18 years) who are admitted to the hospital with a lung infection.

Groups:

LUS Group: These patients will have a lung ultrasound within 24 hours of enrollment. The results will help guide decisions about when to stop antibiotics.

Standard Care Group: These patients will receive regular hospital care, which may include chest X-rays and other tests to guide their treatment.

What Will Be Measured?

Primary Goal: The study will measure how long children and teens stay on antibiotics. The investigators are testing whether LUS can help shorten this time without affecting their recovery.

Secondary Goals: Investigators will also look at how long patients stay in the hospital, whether they need further treatment or care after leaving.

Why is This Important? If this study shows that LUS can safely reduce the use of antibiotics, it could change how doctors treat lung infections in children. Reducing unnecessary antibiotic use can help fight antibiotic resistance and protect children from side effects of unnecessary treatments.

DETAILED DESCRIPTION:
The PLUS-AP Trial (Pediatric Lung Ultrasound to Guide Antibiotic Prescriptions for Hospitalized Children and Adolescents with Lower Respiratory Tract Infections) is a randomized controlled trial designed to assess the effect of pediatric lung ultrasound (LUS) on antibiotic prescribing practices for children and adolescents hospitalized with lower respiratory tract infections (LRTIs). This study aims to explore whether incorporating LUS into clinical decision-making can reduce the unnecessary use of antibiotics without compromising patient care.

Background:

Antibiotics are frequently overprescribed for LRTIs in pediatric populations, contributing to antibiotic resistance and unnecessary adverse events. While chest X-rays are commonly used to diagnose LRTIs, they can be resource-intensive and involve radiation exposure. Lung ultrasound (LUS) is a non-invasive, radiation-free imaging modality that has gained recognition for its utility in diagnosing and monitoring respiratory diseases. This trial will evaluate whether LUS can assist clinicians in making more accurate diagnostic decisions and potentially reduce the use of antibiotics in hospitalized pediatric patients with LRTIs.

Study Objectives:

Primary Objective: To assess whether the use of pediatric lung ultrasound (LUS) reduces the duration of antibiotic treatment in hospitalized children and adolescents diagnosed with LRTIs.

Secondary Objectives:

To evaluate the impact of LUS on the length of hospital stay. To compare clinical outcomes such as the need for escalation to invasive respiratory support, mortality, and readmission rates between the LUS and standard care groups.

To assess the cost-effectiveness of LUS implementation in managing pediatric LRTIs.

Study Design:

The PLUS-AP trial is designed as a phase III, randomized, controlled, patient blinded, single center superiority trial with two parallel groups and a primary endpoint of antibiotic prescriptions by the day of discharge from the hospital. Randomization will be performed as permuted block randomization with a 1:1 allocation.

LUS Group: Participants will undergo lung ultrasound within 24 hours of enrollment, and the results will be used to guide antibiotic therapy decisions, including the duration of antibiotic treatment.

Standard Care Group: Participants will receive standard care, which includes clinical evaluation and any other diagnostic tests, such as chest X-ray, as deemed necessary by the treating physician.

Study Population:

Inclusion Criteria:

* Age between 3 months and 17 years old inclusive
* Currently admitted to the pediatric Ward or boarding in the Emergency Department within 24 hours of admission order due to lower respiratory tract infections.

Exclusion Criteria:

* Sickle cell disease (SCD).
* On chemotherapy or any other immunosuppressive therapy except systemic corticosteroids use of ≤ 5 days duration.
* Cystic fibrosis and other chronic lung diseases except asthma
* Pre-existing and/or congenital neurologic, metabolic, and cardiac conditions
* Hospitalized within the previous month
* Patients with suspected foreign body aspiration -Received antibiotic therapy within the previous week
* Patients admitted under PI's care

Study Interventions:

Lung Ultrasound (LUS): The ultrasound will be exclusively performed by the principal investigator (A.I.), who has credentialing in LUS with more than 4 years of experience, and will be blinded to CXR results. It will take less than 15 minutes, with follow-up scans conducted within 48 hours or prior to discharge to monitor disease progression.

Standard Care: The control group will follow typical hospital procedures, with diagnosis and treatment guided by clinical examination and routine diagnostic tests such as chest X-ray.

Outcome Measures:

Primary Outcome: investigate the effect of adding LUS to standard care on the endpoint of antibiotic prescriptions upon discharge in children hospitalized with LRTIs, compared to standard care and SLUS.

Secondary Outcomes:

To investigate the effect of adding LUS to standard care, as compared to standard care with SLUS, on the end points of:

Trial design

* Length of stay in the hospital
* Rate of complications by 4 weeks after enrollment: admission to ICU, chest tube insertion, mortality
* Frequency of CXR performance within 4 weeks of enrollment
* Rate of antibiotic intake assessed 4 weeks after enrollment
* Rate of hospital readmission within 4 weeks of enrollment.

Expected Impact:

The results of this trial could potentially change clinical practices by providing evidence supporting the use of LUS in reducing unnecessary antibiotic use, thereby reducing the burden of antibiotic resistance in pediatric populations. It could also contribute to the safe and more efficient management of LRTIs in hospitalized children and adolescents.

Estimated Study Timeline:

Study Start Date: april 2025 Study Completion Date: noveber 2026

Sponsor and Investigators:

Principal Investigator: Dr. Ali Ismail Co-Investigators: Dr. Marianne Majdalani, Dr. Jihane Moukhaiber, and others.

ELIGIBILITY:
Inclusion Criteria:

* Age between 3 months and 17 years old inclusive
* Currently admitted to the pediatric Ward or boarding in the Emergency Department within 24 hours of admission order due to lower respiratory tract infections.

Exclusion Criteria:

* Sickle cell disease (SCD).
* On chemotherapy or any other immunosuppressive therapy except systemic corticosteroids use of ≤ 5 days duration.
* Cystic fibrosis and other chronic lung diseases except asthma
* Pre-existing and/or congenital neurologic, metabolic, and cardiac conditions
* Hospitalized within the previous month
* Patients with suspected foreign body aspiration -Received antibiotic therapy within the previous week
* Patients admitted under PI's care

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 176 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Antibiotic Prescription Rate Upon Discharge | Upon discharge (up to 30 days).
  The primary outcome is the rate of antibiotic prescriptions at the time of discharge. This will compare the proportion of children and adolescents with lower respiratory tract infections (LRTIs) who are prescribed antibiotics upon discharge in the experimental group (Lung Ultrasound [LUS]) versus the control group (Sham Lung Ultrasound [SLUS]) or standard care. The aim is to assess whether the use of LUS can reduce unnecessary antibiotic prescriptions at discharge.

DOCUMENTS (1):
  • Study Protocol (2025-02-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT06876766/Prot_000.pdf